CLINICAL TRIAL: NCT07013708
Title: Effectiveness of Low-intensity Laser on Pain in Patients With Supraspinatus Tendinopathy: Randomized Controlled Clinical Trial.
Brief Title: Effectiveness of Low-intensity Laser on Pain in Patients With Supraspinatus Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/06/2024
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Tendinopathy; Pain
Keywords: shoulder; laser; placebo; Tendinopathy
MeSH Terms: conditions — Tendinopathy; Pain | interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator
Masking Description: simple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser treatment (Experimental): Patients diagnosed with laser-treated supraspinatus tendinopathy
  Interventions: Device: Laser
- Placebo Group (Active Comparator): Patients diagnosed with supraspinatus tendinopathy treated with placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Laser — High frequency laser device
  Arms: Laser treatment
Other: Placebo — Same device but without pressing the ON button
  Arms: Placebo Group

SUMMARY:
Tendinopathy is an inflammatory process that occurs in and around the tendon when both are affected by a certain injury. In the case of the supraspinatus muscle it is one of the most frequent causes of shoulder pain. To test the efficacy of laser treatment in reducing shoulder pain caused by supraspinatus muscle tendinopathy. A randomized controlled clinical trial was carried out in which a physiotherapy intervention was performed using therapeutic laser for four weeks, to observe the influence on the pain generated by supraspinatus muscle tendinopathy in the shoulder. A sample of 82 patients was recruited and randomly divided into two groups: experimental group and control group. Laser therapy was applied to the first group and to the second group it was applied as a placebo

ELIGIBILITY:
Inclusion Criteria:

* Age 30-65 years.
* Present a 3 or higher on the visual analogue scale in the shoulder.
* Adequate cognitive capacity for comprehension.
* Tendinopathy of the rotator cuff confirmed by ultrasound at the study center, either by inflammation of the tendon, presence of hypoechoic zones, calcification, fibrillar disorganization and/or neovascularization in the supraspinatus muscle.
* Pain in the proximal side of the arm that is aggravated by abduction.

Exclusion Criteria:

* Laser-specific contraindications (e.g., tumors, presence of pacemaker or defibrillator, pregnancy, etc.).
* History of glenohumeral fracture and rheumatoid arthritis.
* Rheumatic, neurological or structural polymyalgia affecting the joint.
* Previous surgeries.
* Pregnant or breastfeeding women.
* Taking anticoagulants or antiaggregants.
* Diabetes mellitus.
* Cardiac dysfunctions.
* Infiltrative and/or rehabilitative treatment in the two months prior to recruitment.
* Pre-existing diseases associated with pain in the upper extremities.
* Difficulties of follow-up.
* Depression.
* Treatment with another intervention, during the development of the study will not be able to perform.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-05-24 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 12 weeks
  pain scale where 0 is the lowest possible pain score and 10 is the maximum possible pain score

SECONDARY OUTCOMES:
Range of movement | 12 weeks
  joint mobility of the shoulder measured by digital goniometer
pain threshold | 12 weeks
  pressure pain threshold measured by digital algometre

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pontificia de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] So BCL, Lau SCT, Kwok WY, Tse DHT, Man SS. Investigating The Association Between Supraspinatus Tendon Abnormality, Shoulder Pain and Isokinetic Strength in Elite Swimmers: A Cross-Sectional Study. J Sports Sci Med. 2023 Mar 1;22(1):17-27. doi: 10.52082/jssm.2023.17. eCollection 2023 Mar. PMID 36876175
- [Result] Rodeo SA, Nguyen JT, Cavanaugh JT, Patel Y, Adler RS. Clinical and Ultrasonographic Evaluations of the Shoulders of Elite Swimmers. Am J Sports Med. 2016 Dec;44(12):3214-3221. doi: 10.1177/0363546516657823. Epub 2016 Aug 9. PMID 27507844
- [Result] Blevins FT. Rotator cuff pathology in athletes. Sports Med. 1997 Sep;24(3):205-20. doi: 10.2165/00007256-199724030-00009. PMID 9327536
- [Result] Lewis JS. Rotator cuff tendinopathy: a model for the continuum of pathology and related management. Br J Sports Med. 2010 Oct;44(13):918-23. doi: 10.1136/bjsm.2008.054817. Epub 2009 Apr 12. PMID 19364757
- [Result] Haslerud S, Magnussen LH, Joensen J, Lopes-Martins RA, Bjordal JM. The efficacy of low-level laser therapy for shoulder tendinopathy: a systematic review and meta-analysis of randomized controlled trials. Physiother Res Int. 2015 Jun;20(2):108-25. doi: 10.1002/pri.1606. Epub 2014 Dec 2. PMID 25450903
- [Result] Tumilty S, Munn J, McDonough S, Hurley DA, Basford JR, Baxter GD. Low level laser treatment of tendinopathy: a systematic review with meta-analysis. Photomed Laser Surg. 2010 Feb;28(1):3-16. doi: 10.1089/pho.2008.2470. PMID 19708800
- [Result] Notarnicola A, Covelli I, Macchiarola D, Bianchi FP, Cassano GD, Moretti B. The Efficacy of Temperature-Controlled High-Energy Polymodal Laser Therapy in Tendinopathy of the Shoulder. J Clin Med. 2023 Mar 29;12(7):2583. doi: 10.3390/jcm12072583. PMID 37048665
- [Result] Elsodany AM, Alayat MSM, Ali MME, Khaprani HM. Long-Term Effect of Pulsed Nd:YAG Laser in the Treatment of Patients with Rotator Cuff Tendinopathy: A Randomized Controlled Trial. Photomed Laser Surg. 2018 Sep;36(9):506-513. doi: 10.1089/pho.2018.4476. PMID 30188253